CLINICAL TRIAL: NCT05624268
Title: A Phase III, Multicentre, Randomised, Double-blind, Placebo-controlled Study to Investigate the Efficacy, Safety, and Tolerability of COMP360 in Participants With Treatment-resistant Depression
Brief Title: Efficacy, Safety, and Tolerability of COMP360 in Participants With TRD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: COMPASS Pathways (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COMP 005
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 25 mg COMP360 Psilocybin (Experimental): 25 mg COMP360 Psilocybin
  Interventions: Drug: Psilocybin
- Placebo (Placebo Comparator): Matched placebo
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — COMP360 Psilocybin administered under supportive conditions
  Other Names: COMP360

SUMMARY:
Efficacy, Safety, and Tolerability of a single administration of COMP360 in participants with treatment-resistant depression (TRD)

DETAILED DESCRIPTION:
This is a phase III, international, multi-centre, randomised, parallel group, fixed single-dose, double-blind, placebo-controlled study. The study population will include participants aged ≥18 years with TRD.

Overall, 255 participants will be randomised in a 2:1 ratio to receive COMP360 25 mg or placebo.

The study comprises three parts (A, B, and C) and will last approximately 62 weeks including a three- to ten-week Screening Period.

Part A will include a six-week follow-up from initial investigational product (IP) administration.

In this study, the primary aim is to assess the efficacy and safety of a single dose of COMP360 25 mg versus placebo for reducing symptom severity in TRD, when administered with psychological support. This will be assessed in a 6-week, single-dose, double-blind, placebo-controlled part of the study (Part A). Durability of efficacy and long-term safety, and the efficacy and safety of re-treatment will be assessed in a 20-week single-dose, double-blind re-treatment part (Part B), and a 26-week open-label treatment part (Part C).

ELIGIBILITY:
Key Inclusion Criteria:

1. Aged ≥18 years at Screening
2. Major depression without psychotic features (single or recurrent episode as informed by the Diagnostic and Statistical Manual of Mental Disorders, 5th edition [DSM-5])
3. If the current major depressive episode is the participant's first lifetime episode of depression, the length of the current episode must be ≥3 months and ≤2 years at Screening
4. MADRS total score ≥20 at Screening and Baseline to ensure at least moderate severity of depression
5. TRD, defined as failure to respond to an adequate dose and duration of two, three, or four different pharmacological treatments for the current episode as determined through the Massachusetts General Hospital Antidepressant Treatment Response Questionnaire (MGH-ATRQ) and using the supplementary advice on additional antidepressants not included in MGH-ATRQ.
6. At Screening, agreement to discontinue all prohibited medications.

Key Exclusion Criteria:

Psychiatric Exclusion Criteria:

1. Prior or ongoing bipolar disorder, any psychotic disorder, including schizophrenia, schizophreniform disorder, schizoaffective disorder, brief psychotic disorder (unless substance induced or due to a medical condition), antisocial personality disorder as assessed by a structured clinical interview (MINI 7.0.2)
2. Lifetime paranoid, schizoid, schizotypal, histrionic, narcissistic personality disorder, or any ongoing serious psychiatric comorbidity based on medical history and clinical judgement
3. Borderline personality disorder as demonstrated by medical history or the Mini International Neuropsychiatric Interview Plus (MINI plus) - borderline personality disorder module
4. Ongoing post-traumatic stress disorder, obsessive-compulsive disorder, or anorexia nervosa as assessed by medical history and a structured clinical interview (MINI 7.0.2)
5. Psychiatric inpatient within the past 12 months prior to Screening
6. Use of electroconvulsive therapy, deep brain stimulation, or vagus nerve stimulation during the current depressive episode
7. Transcranial magnetic stimulation within the past six months prior to Screening
8. Current enrolment in a psychological therapy programme that will not remain stable for the duration of the study. Psychological therapies cannot have been initiated within 30 days prior to Screening
9. Exposure to COMP360 psilocybin therapy prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
COMP360 25 mg versus placebo for the change from baseline in MADRS total score | Week 6
  Montgomery-Åsberg Depression Rating Scale (MADRS) is a 10-item clinician rated scale measuring depression severity

SECONDARY OUTCOMES:
COMP360 25 mg versus placebo for the change from baseline in SDS total score | Week 6
  Sheehan Disability Scale (SDS) is a brief, five-item self report inventory that assesses functional impairment in work/school, social life, and family life.

CONTACTS AND LOCATIONS:
Locations (40):
- United States (40):
  - University of Arizona College of Medicine - Tuscon, Tucson, Arizona
  - ProScience Research Group, Culver City, California
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Kadima Neuropsychiatry Institute, La Jolla, California
  - University California San Diego, La Jolla, California
  - California Center for Psychedelic Therapy, Los Angeles, California
  - CalNeuro Research Group, Inc, Los Angeles, California
  - Clarity Clinical Research, LLC, Los Angeles, California
  - ATP Clinical Research, Inc., Orange, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Lumos Clinical Research Center, San Jose, California
  - Stanford University, Stanford, California
  - ASCLEPES Research Centers, Thousand Oaks, California
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - Clinical Neurosciecne Solutions, Inc. dba CNS Healthcare, Orlando, Florida
  - APG Research, LLC, Orlando, Florida
  - DMI Health Care Group, Inc, Tampa, Florida
  - Meridien Research/Accel Research, Tampa, Florida
  - Psych Atlanta, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Uptown Research Institute, LLC, Chicago, Illinois
  - Sheppard Pratt Health System, Baltimore, Maryland
  - CBH Health, LLC, Gaithersburg, Maryland
  - Pharmasite Research, Inc, Pikesville, Maryland
  - University of Massachusetts Medical School, North Worcester, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University of Missouri, Columbia, Missouri
  - Midwest Research Group, Saint Charles, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Alivation Research, LLC., Lincoln, Nebraska
  - Bio Behavioral Health, Toms River, New Jersey
  - New York State Psychiatric Institute, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - Insight Clinical Trials, LLC, Beachwood, Ohio
  - Neuro-Behaviroral Clinical Research, Inc., North Canton, Ohio
  - Rivus Wellness & Research Institute, Oklahoma City, Oklahoma
  - Global Medical Institutes, LLC, Scranton Medical Institute, Moosic, Pennsylvania
  - UT Health Science Center at Houston (UTHSC-H), Houston, Texas
  - Cedar Clinical Research, Draper, Utah
  - Core Clinical Research, Everett, Washington

IPD SHARING:
Plan to Share IPD: Undecided